CLINICAL TRIAL: NCT02202395
Title: A Radomized, Double-blind, and Placebo-controlled Multicenter Clinical Trial of Hydroxytriptolide, in Active Rheumatoid Arthritis Patients With an Inadequate Response to Methotrexate
Brief Title: Hydroxytriptolide in Active Rheumatoid Arthritis Patients With an Inadequate Response to Methotrexate
Acronym: T8
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LTS-201-P1.0
Record Dates: First submitted 2014-07-23; First posted 2014-07-29 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Hydroxytriptolide; Rheumatoid Arthritis; Methotrexate; T8; LTS
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 0.25mg (Active Comparator): LTS 0.25mg,qd MTX qw
  Interventions: Drug: LTS 0.25mg
- 0.5mg (Active Comparator): LTS 0.5mg, qd MTX qw
  Interventions: Drug: LTS 0.5mg
- 1.0mg (Active Comparator): LTS 1.0mg,qd MTX qw
  Interventions: Drug: LTS 1.0mg
- Placebo (Placebo Comparator): Placebo qd MTX qw
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LTS 0.25mg — use LTS 0.25mg/d
  Other Names: Hydroxytriptolide
  Arms: 0.25mg
Drug: LTS 0.5mg — use LTS 0.5mg/d
  Other Names: Hydroxytriptolide
  Arms: 0.5mg
Drug: LTS 1.0mg — use LTS 1.0mg/d
  Other Names: Hydroxytriptolide
  Arms: 1.0mg
Drug: Placebo — use placebo once daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of Hydroxytriptolide(LTS) in active rheumatoid arthritis patients with an inadequate response to methotrexate.

DETAILED DESCRIPTION:
1. Investigate the efficacy of Hydroxytriptolide in active RA patients
2. Investigate the safety of Hydroxytriptolide in active RA patients. Especially in female reproductive system.
3. Population PK study.

ELIGIBILITY:
Inclusion Criteria:

* 35-65 years old, female, postmenopausal, parous, nulliparous with no fertility requirements
* 1987 ACR Diagnostic criteria or 2009 ACR/EULAR Diagnostic criteria. X ray of Evaluable Joint in phase I/II/III, Joint Function in Phase I/II/III
* Active RA
* Continuously taking MTX for at least three months, ≥7.5mg/week. Before first study dose, keep in stable MTX dose for at least 4 weeks
* Keep in stable NSAIDs dose or low-dose glucocorticoids for at least 4 weeks before first study dose
* Using non-prohibited combination therapy, keep in stable dose for at least 7 days before first study dose
* Using DMARD should have appropriate withdrawal period:

  * Withdrawal for 4 weeks: Sulfasalazine, Azathioprine, Chloroquine, *Hydroxychloroquine, Auranofin, Penicillamine, Traditional Chinese medicine preparation(TGP, Sinomenine)
  * Withdrawal for 8 weeks: Leflunomide
  * Withdrawal for 8 weeks: Intramuscular, intravenous, intra-articular injection glucocorticoids
* Women with fertility, negative in pregnancy test, and agreed to take contraceptive measures physical
* Voluntary informed consent
* Willing to follow the required regimen and schedule, follow-up examination

Exclusion Criteria:

1. Currently suffering or have suffered from other inflammatory joint diseases, such as mixed connective tissue disease, scleroderma, systemic lupus erythematosus, ankylosing spondylitis, psoriatic arthritis, Reiter's syndrome, bone arthritis, rheumatoid arthritis, gouty arthritis, diagnosis of arthritis before 16yrs
2. With severe non-articular manifestations such as high fever, interstitial pneumonia, pleurisy, pericarditis, severe vasculitis, neuropathy, etc.
3. The evaluable joint underwent the surgical treatment within 2 months
4. Currently or recent have serious, or progression, or disease history not controled, including: liver, kidney, blood, gastrointestinal, endocrine, metabolic, respiratory, cardiovascular, nervous system diseases
5. Currently or have malignancy, lymphoproliferative disease history
6. Continuously use Tripterygium preparations for more than three months and have no effect
7. History of using TNF-a inhibitors of biological agents.(Adalimumab, infliximab, etanercept)
8. Severe or persistent infection within 3 months
9. X-ray shows active pulmonary infection
10. HBV, HCV, HIV, AIDS
11. WBC<4.0×10^9/L, PLT<100×10^9/L, Hb<85g/L
12. AST>2×ULN, ALT>2×ULN
13. Cr>135umol/L
14. Used oral contraceptive druds within 3 months
15. Pregnancy test was positive or lactating patients or patients with birth preparation
16. Have to use the prohibited drugs
17. With clinical symptoms of a serious history of drug abuse or alcohol abuse
18. History of any durg clinical trials within 3 months
19. Allergy to tripterygium
20. Other reasons depends by the investigator

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-06; Primary Completion 2015-04-30 (Actual); Study Completion 2016-12-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline in ACR 20 at 12 weeks and at 24 weeks | 12weeks, 24weeks

SECONDARY OUTCOMES:
Change from baseline in DAS 28 at 12 weeks and at 24 weeks | 12weeks, 24weeks
The proportion of patients reached ACR50 at 12 weeks and 24 weeks | 12weeks, 24weeks
The proportion of patients reached ACR70 at 12weeks and 24weeks | 12weeks,24weeks
Change from baseline in swollen joint count at 12 weeks and 24 weeks | 12weeks,24weeks
Change from baseline in tender joint count at 12weeks and 24weeks | 12weeks,24weeks
Change from baseline in the duration of morning stiffness at 12 weeks and 24 weeks | 12 weeks and 24 weeks
Change from baseline in rest pain at 12 weeks and 24 weeks | 12weeks,24weeks
Change from baseline in PtGA patient global assessment at 12 weeks and 24 weeks | 12 weeks and 24 weeks
Change from baseline in PGA physician global assessment at 12 weeks and 24 weeks | 12 weeks and 24 weeks
Change from baseline in HAQ health assessment questionnaire at 12 weeks and 24 weeks | 12 weeks, 24 weeks
Change from baseline in CRP,ESR,RF,CCP at 12 weeks and 24 weeks | 12 weeks, 24 weeks
Change from baseline in IgA, IgG, IgM at 12 weeks and 24 weeks | 12 weeks, 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chunde Bao, MD, Principal Investigator — Shanghai Jiaotong University School of Medicine, Renji Hospital Ethics Committee
Locations (5):
- China (5):
  - The first affiliated hospital of bengbu medical college, Bengbu, Anhui
  - Changzheng Hospital, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Jiaotong University School of Medicine, Renji Hospital Ethics Committee, Shanghai, Shanghai Municipality
  - Changhai Hospital, Shanghai, Shanghai Municipality